CLINICAL TRIAL: NCT04870203
Title: Combination of Baricitinib and Anti-TNF vs. Baricitinib in Patients With Rheumatoid Arthritis: a Randomized Controlled Phase III Trial
Brief Title: Combination of Baricitinib and Anti-TNF in Rheumatoid Arthritis
Acronym: CRI-RA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Eli Lilly and Company (Industry); Biogen (Industry); Ministry for Health and Solidarity, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHUBX 2019/56
Record Dates: First submitted 2021-04-26; First posted 2021-05-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
Keywords: baricitinib; adalimumab; etanercept; placebo
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Period A : placebo-controlled trial *** Period B : controlled trial - study switch to an open-label design from the 17th August 2024
Who Masked: Participant, Care Provider, Investigator
Masking Description: Period A : Participant / Care provider / Investigator *** Period B : An independent efficacy assessor will perform the joint evaluation, whereas the investigator will evaluate safety.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Period A : baricitinib + anti-TNF (Experimental)
  Interventions: Drug: baricitinib treatment; Drug: anti-TNF therapy
- Period A : baricitinib + placebo (Placebo Comparator)
  Interventions: Drug: baricitinib treatment; Drug: Placebo
- Period B : baricitinib + anti-TNF (Experimental)
  Interventions: Drug: baricitinib treatment; Drug: anti-TNF therapy
- Period B : baricitinib (Active Comparator)
  Interventions: Drug: baricitinib treatment

INTERVENTIONS:
Drug: baricitinib treatment — 4 mg daily during 12 months
Drug: anti-TNF therapy — adalimumab at 40 mg every 2 weeks or etanercept 50 mg per week according to treatments history
  Arms: Period A : baricitinib + anti-TNF; Period B : baricitinib + anti-TNF
Drug: Placebo — 40 mg every 2 weeks during 6 months only during Period A
  Arms: Period A : baricitinib + placebo

SUMMARY:
As stated by the European League Against Rheumatism (EULAR) and the Société Française de Rhumatologie (SFR), treatment of patients with rheumatoid arthritis (RA) should target sustained remission or at least low disease activity. However, despite significant advances based on various combinations of conventional synthetic disease-modifying antirheumatic drugs (DMARDs) and biologic DMARDs, RA therapies meet treatment goals only in some patients:

* 40 to 50% of patients with early RA, treated with methotrexate (MTX) monotherapy as first-line therapy,
* 20 to 30% of patients treated with a combination of MTX and biologic as second-line therapy.
* Less than 10% of patients treated with a combination of MTX and another targeted DMARD, such as baricitinib, as third-line therapy.

Therefore, new strategies targeted at achieving a higher percentage of remission are needed, that do not require waiting for multiple failed therapies. Combinations of biologics have shown synergistic improvement of symptoms in murine models of RA relative to the improvement observed with either agent alone. However, in RA patients, only five randomised clinical trials (RCTs) have explored the efficacy and safety of combining tumour necrosis factor (TNF) inhibitor with another biologic (anakinra, abatacept, rituximab or bimekizumab).

Baricitinib is a selective, reversible and competitive inhibitor of Janus kinases (Jaki). This treatment is efficient in a number of therapeutic scenarios in RA and showed a clinical superiority over adalimumab in one RCT (RA-BEAM study in MTX inadequate responders). Of note, baricitinib inhibits many of the pro-inflammatory cytokines involved in the pathogenesis of RA but does not block signalling downstream of TNF. Owing to the interest in combining different mechanisms of action, the investigators plan to assess the efficacy and safety of combination therapy with baricitinib and a TNF inhibitor. The investigators are aware that combining targeted therapies is not recommended due to a potential increase in the frequency of serious adverse events. However, several case series on patients treated with a combination of targeted therapies have been published, suggesting a certain efficacy in patients with refractory RA. The first ones focused on inflammatory bowel diseases and psoriasis, but more recently, combination of tofacitinib (which belongs to the same Jaki family as baricitinib) with various biologics has been reported in a sample of RA patients. No serious adverse effects were reported over a mean of approximately 11 months of therapy. The clinical improvement was mild but noticeable in these refractory RA cases.

Recently, data of interest from the RA-BEAM study have been reported. Patients who switched from adalimumab to baricitinib showed improvements in disease control. Because the switch from adalimumab to baricitinib occurred without a washout period, and because adalimumab has a mean circulating half-life of approximately 14 days, patients would have received several weeks of dual TNF and Jak1/Jak2 inhibition in the course of the change of treatment. The observation of increased efficacy, with no apparent acute safety issues during the weeks when patients were exposed to both adalimumab and baricitinib, is of interest, and supports our strategy to combine the two treatments for patients with refractory RA.

The investigators consider that there is a need for investigation into the addition of anti-TNF to baricitinib in patients suffering of refractory RA (inadequate response to TNF inhibitors). The investigators hypothesize that in this population, based on ACR50 score, this combination therapy will decrease disease activity more efficiently than a switch to another targeted DMARD, such as baricitinib.

DETAILED DESCRIPTION:
Intensive combination therapies have revolutionised the management of solid neoplasms, hematologic malignancies, and acquired-immune-deficiency syndrome. These intensive strategies are based on the need to obtain rapid control of disease activity to afford the chance of stable full remission and avoid irreversible complications. The same goal applies to management of RA. Because current therapeutic strategies may fall short of these target goals and fail to improve quality of life in some patients, novel approaches are needed to improve outcomes. RA is a complex disease involving numerous cell types and inflammatory mediators of innate and adaptive immune systems. The investigators are aware that most of combination bDMARD strategies have been associated with little or no incremental benefit in efficacy compared to single-biologic therapy. However, our study will target mechanisms that differ from those in previous studies. Strategies that simultaneously target different pathways involved in the pathogenesis of RA may enhance treatment responses in patients with RA. Of note, baricitinib does not directly block signalling downstream of TNF, even if an indirect effect on TNF production is likely to occur. Targeting multiple inflammatory cytokines in combination may lead to more effective treatment and enhanced clinical responses in patients with RA compared to the current second-line strategies. The different mechanisms of action of baricitinib and anti-TNF, should ensure the efficacy of the combination. No concurrent trial evaluating similar strategies is registered at ClinicalTrial.gov.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Age between 18 and 65 years-old;
* Adult patient with a diagnosis of RA as defined by the ACR/EULAR 2010 criteria for the classification of RA;
* Patient who presents an inadequate response to at least one bDMARD or tsDMARD for at least 12 weeks prior to study entry at a dose that is considered acceptable to assess clinical response adequately;
* Patient affected by active RA (DAS28-ESR > 3.2 or sDAI > 11 or cDAI > 10) eligible to receive a bDMARD or tsDMARD according to the French Society of Rheumatology guidelines;
* Patient treated by prednisone dosage ≤ 10mg per day. The corticosteroids dosage will be decreased to 7,5 mg/day at the beginning of the study (W0);
* Person affiliated with or beneficiary of the French social security scheme;
* Free, informed and written consent signed by the participant and the investigator (on the day of inclusion at the latest and before any examination required by the research project).

Exclusion Criteria:

* Patient previously treated with baricitinib;
* Patient previously treated by both adalimumab and etanercept. If the patient received previously only one of these two treatments, he/she can be included in the study with the treatment he/she has not yet received (if he/she is randomized in the experimental COMBI group);
* Patient affected by another form of inflammatory arthritis with the exception of secondary Sjögren syndrome;
* Patient who presents contraindications to the study treatments;
* Patients who is an active smoker or former smokers with a maximum exposure of 10 years;
* Patient who is currently receiving glucocorticosteroids at doses >10 mg of prednisone per day (or equivalent) or has been receiving an unstable dosing regimen of corticosteroids within 4 weeks of study entry;
* Patient who is currently receiving more than 1 concomitant csDMARD (MTX, leflunomide, hydroxychloroquine or sulfasalazine) at the time of study entry;
* Patient who is currently receiving or has received csDMARDs (eg, gold salts, cyclosporine, azathioprine, or any other immunosuppressives) other than MTX (up to 25 mg/week), leflunomide (up to 20 mg/day), hydroxychloroquine (up to 400 mg/day), or sulfasalazine (up to 3000 mg/day) within 4 weeks prior to study entry.
* Doses of hydroxychloroquine or sulfasalazine should be stable for at least 4 weeks prior to study entry; if either has been recently discontinued, the patient must not have taken any dose within 4 weeks prior to study entry.
* Immunosuppression related to organ transplantation is not permitted;
* Patient who has received any parenteral corticosteroid administered by intramuscular or intravenous injection within 4 weeks prior to study entry, or is anticipated to require parenteral injection of corticosteroids during the study;
* Patient who had 3 or more joints injected with intraarticular corticosteroids or hyaluronic acid within 4 weeks prior to study entry. Joints injected with intraarticular corticosteroids or hyaluronic acid within 2 weeks prior to study entry or within 6 weeks prior to planned randomization cannot be counted in the TJC and SJC for entry or enrollment purposes;
* Patient with haemoglobin less than 80 g/L, absolute lymphocyte count lower than 0.5×109/L, absolute neutrophil count less than 1×109/L, or platelet count less than 100×109/L; clearance creatinine less than 60 mL/min; total bilirubin more than 1.5 times the upper limit of normal (ULN) at screening, aspartate aminotransferase, or alanine amino-transferase more than 2 times the upper limit of normal (ULN) at screening.
* Patient with co-administration with OAT3 inhibitors (such as probenecid);
* Patient who has a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric diseases or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute a risk when taking investigational product or could interfere with the interpretation of data;
* Patient with an history of Moderate to severe heart failure (NYHA classes III/IV);
* Patient with an history of Major Adverse Cardiovascular Events (non-fatal myocardial infarction or non-fatal stroke);
* Patient who has a history of Venous Thromboembolic Event (VTE) (DVT/PE) within 12 weeks prior to randomization or have a history of recurrent (>1) VTE (DVT/PE). Prior DVT with PE where events overlapped in time (i.e., with PE considered resulting from DVT) is not considered recurrent DVT/PE for the purpose of this criterion.
* Patient who has been exposed to a live vaccine within 12 weeks prior to planned randomization or are expected to need/receive a live vaccine during the course of the study (with the exception of herpes zoster vaccination). Investigators should review the vaccination status of their patients and follow the local guidelines for adult vaccination with nonlive vaccines intended to prevent infectious disease prior to entering patients into the study;
* Patient with an active cancer;
* Patient with malignancy or history of malignancy;
* Patient who has a current or recent (<30 days prior to study entry) clinically serious viral, bacterial, fungal, or parasitic infection;
* Patient who is immunocompromised and, in the opinion of the investigator, is at an unacceptable risk for participating in the study;
* Patient with a history of active hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV);
* Patient who had household contact with a person with active tuberculosis (TB) and did not receive appropriate and documented prophylaxis for TB;
* Patient who has evidence of active TB or has previously had evidence of active TB and did not receive appropriate and documented treatment;
* Patient who has evidence of latent TB (as documented by a positive Purified Protein Derivative (PPD), no clinical symptoms consistent with active TB, and a normal chest x-ray at screening) unless patient completes at least 3 weeks of appropriate treatment prior to study entry and agrees to complete the remainder of treatment while in the trial
* Patient who had any major surgery within 8 weeks prior to study entry or will require major surgery during the study that, in the opinion of the investigator, would pose an unacceptable risk to the patient;
* Pregnant or breastfeeding woman, or woman who refuses to use an effective contraception during the study course;
* Patient governed by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieve an ACR 50 response | At weeks 24 after baseline
  in each treatment group (COMBI group (anti-TNF therapy + baricitinib) vs. MONO group (baricitinib conventional therapy)).
Quantitative change in DAS28-CRP | At weeks 24 after baseline
  in each treatment group (COMBI group (anti-TNF therapy + baricitinib) vs. MONO group (baricitinib conventional therapy)).

SECONDARY OUTCOMES:
Proportion of adverse events (AE) and serious adverse events (SAE) in each treatment group | weeks 52 after baseline (Day 0)
Proportion of patients who achieve an ACR20 response in each treatment group | At weeks 4, 12 and 24 after baseline (Day 0)
Proportion of patients who achieve an ACR70 response in each treatment group | At weeks 4, 12 and 24 after baseline (Day 0)
Proportion of patients who achieve an ACR50 response in each treatment group | At weeks 4 and 12 after baseline (Day 0)
Proportion of patients who present a EULAR response according to DAS28-ESR, in each treatment group | at weeks 4, 12 and 24 after baseline (Day 0)
Proportion of patients who achieve remission or low disease activity according to DAS28-ESR in each treatment group | at weeks 4, 12 and 24 after baseline (Day 0)
Quantitative change in DAS28-ESR score (Disease Activity Score on 28 joints using Erythrocyte Sedimentation Rate) in each treatment group of treatment, varying from 0 to 9.55 with higher score means worse outcome. | between baseline and each visit (until week 24 included)
Quantitative change in DAS28-CRP score between baseline and each visit (until week 24 included) in each treatment group of treatment, varying from 0.96 to 9.04 with higher score means worse outcome. | between baseline and each visit (until week 24 included)
  Disease Activity Score on 28 joints using C-Reactive Protein level (DAS28-CRP)
Quantitative change in sDAI score (simplified Disease Activity Index) between baseline and each visit (until week 24 included) in each treatment group of treatment, varying from 0 to 100 with higher score means worse outcome. | between baseline and each visit (until week 24 included)
Quantitative change in cDAI score (clinical Disease Activity Index) between baseline and each visit (until week 24 included) in each treatment group of treatment, varying from 0 to 76 with higher score means worse outcome. | between baseline and each visit (until week 24 included)
Proportion of patients who decrease the glucocorticosteroid dose ≤ 5 mg per day, sustained from week 12 to week 24, among patients with a baseline dose > 5 mg per day, in each treatment group. | At baseline (Day 0) and weeks 24 after baseline (Day 0)
Drug retention rates in each treatment group | at weeks 4, 12 and 24 after baseline (Day 0)
Quantitative change in patient-reported outcome in each treatment group Health Assessment Questionnaire (HAQ), varying from 0 to 3 with higher score means worse outcome. | between baseline, weeks 4, 12 and 24 visit
Quantitative change in patient-reported outcome in each treatment group | between baseline, weeks 4, 12 and 24 visit
  Functional Assessment of Chronic Illness Therapy (FACID)
Quantitative change in patient-reported outcome in each treatment group Rheumatoid Arthritis Impact of Disease questionnaire (RAID), varying from 0 to 10 with higher score means worse status. | between baseline, weeks 4, 12 and 24 visit
Proportion of participants maintaining an ACR50 response, remission or low disease activity in each treatment group. | at week 52 after baseline (Day 0)
Quantitative change in DAS28-ESR score (Disease Activity Score on 28 joints using Erythrocyte Sedimentation Rate) in each treatment group, varying from 0 to 9.55 with higher score means worse outcome. | between weeks 24 and 52 after baseline (Day 0)
Quantitative change in DAS28-CRP score (Disease Activity Score on 28 joints using C-Reactive Protein level) in each treatment group, varying from 0.96 to 9.04 with higher score means worse outcome | between weeks 24 and 52 after baseline (Day 0)
Quantitative change in sDAI score (simplified Disease Activity Index) in each treatment group, varying from 0 to 100 with higher score means worse outcome. | between weeks 24 and 52 after baseline (Day 0)
Quantitative change in cDAI score (clinical Disease Activity Index) in each treatment group, varying from 0 to 76 with higher score means worse outcome. | between weeks 24 and 52 after baseline (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe RICHEZ, Prof, Principal Investigator — University Hospital, Bordeaux; Edouard LHOMME, MD, Study Chair — University Hospital, Bordeaux
Locations (36):
- France (35):
  - CH de la Côte Basque - service de rhumatologie, Bayonne
  - CH de Belfort - service de rhumatologie, Belfort
  - AP-HP - Hopital Avicenne - service de rhumatologie, Bobigny
  - CHU de Bordeaux - service de rhumatologie, Bordeaux
  - CHU de Brest - Service de rhumatologie, Brest
  - Clinique de l'Infirmerie - service de rhumatologie, Caluire-et-Cuire
  - CHU de Clermont-Ferrand - service de rhumatologie, Clermont-Ferrand
  - CH de Dax - service de rhumatologie, Dax
  - CHD VENDEE - service de rhumatologie, La Roche-sur-Yon
  - AP-HP - Hôpital Kremlin-Bicêtre - service de rhumatologie, Le Kremlin-Bicêtre
  - CH du Mans - service de rhumatologie, Le Mans
  - CH Emile Roux - service rhumatologie, Le Puy-en-Velay
  - Polyclinique de Limoges - service de rhumatologie, Limoges
  - Groupement des Hôpitaux de l'Institut Catholique de Lille - service de rhumatologie, Lomme
  - AP-HM - service de rhumatologie, Marseille
  - Hôpital Saint-Joseph - service de rhumatologie, Marseille
  - CHU de Montpellier - service de rhumatologie, Montpellier
  - CHU de Nice - service de rhumatologie, Nice
  - CH de Niort - service de rhumatologie, Niort
  - CHU de Nîmes - service de rhumatologie, Nîmes
  - Nouvel Hôpital Orléans La Source - service de rhumatologie, Orléans
  - AP-HP - Hôpital Bichat - service de rhumatologie, Paris
  - AP-HP - Hôpital Cochin - service de rhumatologie, Paris
  - AP-HP - Hôpital La Pitié-Salpetrière - service de rhumatologie, Paris
  - AP-HP - Hôpital Saint-Antoine - service de rhumatologie, Paris
  - CH de Pau - service de rhumatologie, Pau
  - Hospices Civils de Lyon - service de rhumatologie, Pierre-Bénite
  - Hopital NOVO - service de rhumatologie, Pontoise
  - CH de Reims - service de rhumatologie, Reims
  - CHU de Saint-Etienne- service de rhumatologie, Saint-Etienne
  - CH de Saint-Malo - service de rhumatologie, St-Malo
  - CHRU de Strasbourg - service de rhumatologie, Strasbourg
  - CHU de Toulouse - service de rhumatologie, Toulouse
  - CHRU du Tours - service de rhumtologie, Tours
  - CHRU de Nancy - service de rhumatologie, Vandœuvre-lès-Nancy
- service de Rhumatologie - CH Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No